CLINICAL TRIAL: NCT03208777
Title: Telomeric Abnormalities in Benign and Malignant Colorectal Diseases by Fluorescent in Situ Hybridization Technique
Brief Title: Telomeric Abnormalities in Colorectal Diseases by Fluorescent in Situ Hybridization Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, fatma magdy zidan, principle investigator, Assiut University
Other Study IDs: FISH
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Tumor Gastric
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: taking blood samples from apparently healthy people
  Interventions: Genetic: taking blood samples
- benign colorectal: taking blood samples from patients
  Interventions: Genetic: taking blood samples
- malignant colorectal: taking blood samples from patients
  Interventions: Genetic: taking blood samples

INTERVENTIONS:
Genetic: taking blood samples — taking blood samples and measure telomeric abnormalities

SUMMARY:
Colorectal carcinoma is a heterogeneous disease that is caused by the interaction of genetic and environmental factors. colorectal carcinoma encompasses a complex disease with different molecular pathways and biological characteristics arising from a multi-step process that implicates several genetic and epigenetic events . The multi-step genetic model involves the loss of function of tumor suppressor genes, such as adenomatous polyposis coli (APC), Telomeres could be a promising marker due to the fact that their lengths change in the colorectal polyp-carcinoma sequence . Moreover, telomere length (TL) is altered in blood cells in patients with colorectal carcinoma

* These findings could suggest that changes in TL may take place before the development of the tumor .

The two main forms of inflammatory bowel disease (IBD), ulcerative colitis (UC) and Crohn's disease (CD) are characterized by chronic intestinal inflammation and risk of progression to colon cancer. One proposed cause of the latter characteristic is chromosome instability, since the rearrangement of genetic material can lead to activation of oncogenes, loss of tumor suppressor genes and other changes that lead to uncontrolled cell growth. Chromosome instability is particularly associated with UC and has been observed in colon epithelial cells and peripheral blood mononuclear cell. Since genomic instability in peripheral blood mononuclear cells (PBMCs) has been used as a biomarker for global cancer risk in a number of diseases, the latter observation suggests the possibility of a chromosome instability syndrome in UC that could affect all tissues. One possible cause of chromosome instability is telomere dysfunction .

DETAILED DESCRIPTION:
Human chromosomes are capped and stabilized by telomeres, which not only protect them from damage but also have a role in regulating cellular senescence. After reaching a critical length, telomeres experience a double DNA change and cells will eventually enter senescence (replication) or cell death . Telomere length and telomere shortening have been long hypothesized to be a biological marker of aging at the cellular level and a potential mechanism of carcinogenesis. Genomic instability is a critical factor in the initiation and progression of human cancers. One mechanism that underlies genomic instability is loss of telomere function .

fluorescent in situ hybridization is a molecular diagnostic technique that utilizes labeled DNA probes to detect or confirm gene or chromosome abnormalities. fluorescent in situ hybridization is often utilized for both research and diagnosis of hematological malignancies and solid tumors. Conceptually, fluorescent in situ hybridization is a very straightforward technique whereby a DNA probe is hybridized to its complementary sequence on chromosomal preparations previously fixed on microscope slides . fluorescent in situ hybridization is able to detect cells that have chromosomal abnormalities consistent with neoplasia .

There has been a surge of published studies which assessed the association between telomere length and development of colorectal carcinoma. Thus, a meta-analysis addressing colorectal carcinoma and telomere length would be a useful addition to the current information in this area.

ELIGIBILITY:
Inclusion Criteria:

* Adult age group ˃ 18 years.
* Newly diagnosed cases (no previous treatment).
* No treatment was taken for HCV infection.

Exclusion Criteria:

* age group < 18 years.
* Patients with malignancy of other type.
* Patients not diagnosed by endoscopy or biopsy (not surely diagnosed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients with colorectal benign or malignant disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
presence of telomeric abnormalities | one year
  measure percentage of telomeric abnormalities in benign and malignant colorectal diseases

CONTACTS AND LOCATIONS:
Overall Officials: fatma magdy zidan, residant, Principal Investigator — South Egypt Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosman F, Yan P. Molecular pathology of colorectal cancer. Pol J Pathol. 2014 Dec;65(4):257-66. doi: 10.5114/pjp.2014.48094. PMID 25693079